CLINICAL TRIAL: NCT05119348
Title: Transmission of COVID19 in Crowded Environments
Brief Title: Transmission of Coronavirus Disease 2019 (COVID19) in Crowded Environments
Acronym: TRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Desmond Tutu HIV Foundation (Other)
Collaborators: Amsterdam Institute for Global Health and Development (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREC 284 2020
Record Dates: First submitted 2021-11-12; First posted 2021-11-15 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Covid19; Sars-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The study design is a type 2 hybrid cluster (household) randomised controlled trial, with outcomes assessed on index patients and their household contacts. After completing consent, 120 households will be randomised in a 1:1 ratio (60 per arm).
Who Masked: Investigator
Masking Description: The investigators were not made aware of participants study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stop coronavirus (STOPCOV) (Experimental): A fieldworker will deliver the STOPCOV pack and personal protective equipment at baseline. The fieldworker will communicate with intervention households daily, delivering STOPCOV hygiene information.
  Interventions: Other: STOPCOV
- Control (No Intervention): Participants received no additional messaging about managing COVID19 in the household.

INTERVENTIONS:
Other: STOPCOV — Fieldworkers delivered an infection mitigation intervention which consisted of personal protective equipment and messaging on managing COVID19 and reducing onward transmission of SARS-CoV-2 infection.
  Arms: Stop coronavirus (STOPCOV)

SUMMARY:
South Africa recorded it's first coronavirus disease 2019 (COVID19) case on March 5, 2020. In response to the COVID19 outbreak World Health Organisation recommendations, South Africa implemented non-pharmaceutical recommendations. The major risk mitigation factors recommended by World Health Organisation and others - physical distancing and hygiene - are extremely difficult to implement in much of Africa. The investigators will conduct a randomised controlled trial to investigate the effect of an infection mitigation intervention to assess the effect on household transmission of severe acute respiratory syndrome (SARS) coronavirus (CoV) 2 in household settings with an index patient diagnosed SARS-CoV-2 positive.

DETAILED DESCRIPTION:
The major risk mitigation factors recommended by World Health Organisation and others - physical distancing and hygiene - are extremely difficult to implement in much of Africa. Newly diagnosed SARS-CoV-2 index patients will be identified and recruited from a mobile clinic and local community clinics conducting SARS-CoV-2 testing. Index cases and their households will be invited to enroll. The study design is a type 2 hybrid cluster (household) randomised controlled trial, with outcomes assessed on index patients and their household contacts. 120 consecutively newly diagnosed index patients (GeneXpert severe acute respiratory syndrome coronavirus 2 PCR) and up to 6- 8 household contacts will be invited to participate in the trial as part of the prospective observational study evaluating transmission and symptoms. After completing consent, households will be randomised in a 1:1 ratio in blocks of 10 (60 households per group). Klipfontein is a resource-limited, densely populated, high HIV/tuberculosis disease burden areas in Cape Town. Newly diagnosed COVID19 cases will be identified from two sources: screening conducted in Desmond Tutu Health Foundation mobile screening units and local public sector clinics working closely with Desmond Tutu Health Foundation. Consecutive cases (n=120 cases and households) will be invited to participate in the randomised trial and prospective longitudinal follow up of up to 6- 8 household contacts. The contacts will be followed up after informed consent to SARS-CoV-2 screening, symptomatic questionnaires weekly up to 1 month. After enrolment, the household will be randomised to the infection mitigation intervention or enhanced usual care messaging. Baseline demographic, household characteristics questionnaire will be administered, and each household occupant invited to participate. Following consent procedures, household contacts (HHC) will be screened at baseline and weekly for 4 weeks for evidence of COVID19 infection. Specifically, the research team will conduct SARS-CoV-2 GeneXpert PCR testing and antibody serology. They will collate self- administered daily symptom checks on a weekly basis. The investigators will recruit 120 households over 1-11 months. The investigators will initiate a prospective longitudinal follow up of the household contacts of each case for 4 weeks in each case.

The investigators will calculate proportion of SARS-CoV-2 transmission from index cases in each household over 4- week period and describe the proportion of symptomatic and asymptomatic SARS-CoV-2 infection in a high density, low resourced community. Investigate the impact of the infection mitigation intervention by comparing incidence in households randomised to intervention versus standard of care. Secondary outcomes for the trial will include clinical outcomes (hospitalisations, death), linkages to care for people, psychosocial functioning, and stigma.

ELIGIBILITY:
Inclusion Criteria:

* recently diagnosed SARS-CoV-2 positive
* Individual >12 years
* Able to give assent if <18 years with parental/guardian consent
* Able to give consent> 18 years
* Self-isolating at home at the time of COVID diagnosis

Exclusion Criteria:

* <12 years
* Unable to give consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda-Gail Bekker, MBChB, PhD, Principal Investigator — Desmond Tutu Health Foundation
Locations (1):
- Desmond Tutu Health Foundation, Cape Town, WC, South Africa

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data with other researchers.

REFERENCES:
- [Derived] Smith P, Little F, Hermans S, Davies MA, Wood R, Orrell C, Pike C, Peters F, Dube A, Georgeu-Pepper D, Curran R, Fairall L, Bekker LG. A prospective randomised controlled trial investigating household SARS-CoV-2 transmission in a densely populated community in Cape Town, South Africa - the transmission of COVID-19 in crowded environments (TRACE) study. BMC Public Health. 2024 Jul 17;24(1):1924. doi: 10.1186/s12889-024-19462-1. PMID 39020307

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stop Coronavirus (STOPCOV) | Control
Started | 137 | 108
Completed | 137 | 108
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stop Coronavirus (STOPCOV) | Control | Total
Number analyzed (Participants) | 137 | 108 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (16.6) | 39.9 (17.1) | 39.1 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 60 | 139
  Male | 58 | 48 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 69 | 22 | 91
  Race: Coloured | 68 | 82 | 150
  Race: Indian | 0 | 3 | 3
  Race: Prefer not to say | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 137 | 108 | 245

OUTCOME MEASURES:

1. Primary Outcome: SARS-CoV-2 Infection
Description: Number of participants with positive SARS-CoV-2 PCR result
Time Frame: 4 weeks
Population: Number of participants where there was a change observed in their negative to a positive SARS-CoV-2 PCR result
Measure: Count of Participants; unit: Participants
Arm/Group | Stop Coronavirus (STOPCOV) | Control
Number analyzed (Participants) | 137 | 108
Participants | 4 | 2

2. Secondary Outcome: COVID19 Symptoms
Description: Number of participants with SARS-CoV-2 serology antibody positive result
Time Frame: 4 weeks
Population: Number of participants where there was a change observed in their negative to a positive SARS-CoV-2 serology result
Measure: Count of Participants; unit: Participants
Arm/Group | Stop Coronavirus (STOPCOV) | Control
Number analyzed (Participants) | 137 | 108
Participants | 11 | 9

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Stop Coronavirus (STOPCOV) | Control
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/108
Other Adverse Events (participants affected / at risk) | 15/137 | 4/108
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stop Coronavirus (STOPCOV) (N=137) | Control (N=108)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pressure in chest (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Somnolence/ drowsy/ sleepy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Confused/ disoriented (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT05119348/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT05119348/SAP_001.pdf